CLINICAL TRIAL: NCT00257309
Title: TRIANA: A Randomized Trial to Compare the Efficay and Safety of Thrombolysis With Primary Angioplasty as Initial Reperfusion Therapy in Older Patients (>= 75 Years Old) With Acute Myocardial Infarction
Brief Title: Thrombolysis Versus Primary Angioplasty for AMI in Elderly Patients
Acronym: TRIANA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Spanish Society of Cardiology (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); Sanofi (Industry); Cordis US Corp. (Industry); Medtronic (Industry); Guidant Corporation (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Héctor Bueno, (Past) President. WG on IHD, Spanish Society of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT 2004-001943-31; FIS PI042122
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Elderly; Thrombolysis; Primary angioplasty; Randomized trial; Efficacy; Safety
MeSH Terms: interventions — Tenecteplase; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thrombolysis (Active Comparator): Weight adjusted tenecteplase bolus + Unfrationated heparin
  Interventions: Drug: Tenecteplase + UFH (+ clopidogrel, since 01/97)
- Primary angioplasty (Active Comparator): Primary angioplasty
  Interventions: Procedure: Primary angioplasty

INTERVENTIONS:
Drug: Tenecteplase + UFH (+ clopidogrel, since 01/97)
  Arms: Thrombolysis
Procedure: Primary angioplasty
  Arms: Primary angioplasty

SUMMARY:
General objective: To compare the efficacy and safety of primary angioplasty(PA) with that of thrombolytic therapy (TT) for the treatment of AMI in patients >=75 years old with ST-segment elevation or LBBB AMI <6 hours of evolution without contraindications for TT.

Hypothesis: The therapeutical strategy based on PA is superior to that based initially on TT in patients >=75 years old with AMI.

Participating Centers: 27 Spanish hospitals performing >50 PA/year. Primary Endpoint (PE): Incidence of the aggregate of death of any cause, reinfarction or disabling stroke at 30 days. There are also 7 secondary endpoints (SE).

Procedure: Diagnosis of inclusion/exclusion criteria --> Centralized randomization --> Treatment allocation to 1) TT with weight adjusted TNK + unfractionated heparin or 2) PA within 120 minutes. Estimated Sample size and recruitment time: 570 patients in 19 months. Follow-up: Blinded evaluation of events (PROBE regulations) specified in PE and SE at 30 days and 12 months. Quality control: 100% variable and follow-up review by external CRO. Safety Committee and Event Adjudication Committee formed by experts not participating in the study.

DETAILED DESCRIPTION:
Hypothesis of the study. In patients of 75 or more years of age with AMI and ST-elevation or LBBB, the treatment strategy based on primary angioplasty is superior to the treatment strategy based on initial fibrinolytic therapy for reducing the incidence of death, re-infarction and disabling CVA at 30 days. This benefit is maintained at 12 months.

Objectives General objective of the study. To compare the efficacy and safety of primary angioplasty and fibrinolytic treatment in >=75 year-old patients with AMI eligible for fibrinolytic therapy in Spanish medical centers with an active program of primary angioplasty.

Primary end point: Incidence of the combined end point of all-cause death, re-infartion or disabling stroke at 30 days

Secondary end points:

* All-cause death at 30 days
* Incidence of the combined end point of all-cause death, disabling CVA or de novo heart failure at 30 days
* Incidence of recurrent ischemia requiring emergency catheterization in the first 30 days
* Cause of death at 30 days classified in three groups:

  1. Shock or heart (pump) failure
  2. Mechanical complications (ruptures) or electromechanical dissociation
  3. Other causes (including bleeding)
* Incidence of major bleeding during hospital admission
* All-cause mortality at 12 months
* Period of time elapsed until presentation of any of the composite of all-cause death, reinfarction or disabling CVA at 12 months
* Period of time elapsed until the presentation of any composite of all-cause death, reinfarction, disabling CVA or non-elective hospital readmission for cardiac causes (unstable angina, heart failure, non-elective coronary revascularization at 12 months.

TYPE AND DESIGN OF THE CLINICAL TRIAL Clinical trial status Phase IV trial Description of randomization process The treatment strategy will be determined by a centralized randomization process, using a telephone system. Eligible patients will be randomized to one of two (2) treatment arms: fibrinolytic treatment or primary angioplasty.

Control and design This is a randomized multicenter, open blind clinical trial designed to compare the efficacy and safety of primary angioplasty vs. thrombolytic treatment in >=75 year-old patients with AMI and ST-elevation or de novo LBBB, eligible for thrombolysis, admitted at Spanish medical centers that have an active primary angioplasty program, within the first 6 hours after symptom onset.

Masking techniques Being an open trial there are not masking techniques, nor will there be an emergency opening procedure of emergency codes.

Pre-inclusion / clearance period Not applicable

SUBJECT SELECTION Inclusion / exclusion criteria Subjects must be >=75 years of age with AMI and ST-elevation or de novo LBBB, eligible for thrombolytic therapy, admitted in any Spanish medical center in which there is an active primary angioplasty program within the first 6 hours after symptom onset.

Each patient must fulfill all inclusion criteria and none of the exclusion criteria.

Inclusion criteria:

1. Subjects of 75 or more years of age
2. Diagnosis of AMI: chest pain or any symptom of myocardial ischemia of, at least, 20 minutes of duration, not responding to nitrate therapy, an evolution period of less than 6 hours after symptom onset until randomization process, and, at least, one of the following alterations:

   1. ST-elevation >=2 mm in 2 or more precordial leads
   2. ST-elevation >=1 mm in 2 or more anterior leads
   3. Complete de novo (or probably de novo) left bundle branch block (LBBB)
3. Subject should be able to give informed consent prior to randomization process and should agree to fulfill all procedures described in the protocol, including follow-up after hospital discharge. A written consent signed by a close relative with witness is also acceptable.

Exclusion criteria:

1. Documented contraindication to the use of fibrinolytics. 1.1. Internal active bleeding or known history of hemorrhagic diathesis 1.2. History of previous CVA of any kind or at any time 1.3. Intracranial tumor, arteriovenous malformation, aneurysm or cerebral aneurysm repair 1.4. Major surgery, parenchymal biopsy, ocular surgery or severe traumatism in the 6 weeks prior to randomization 1.5. Unexplained puncture in a non-compressible vascular location in the last 24 hours prior to randomization 1.6. Confirmed arterial hypertension with a reliable measurement of systolic AP >180 mmHg or diastolic AP >110 mmHg 1.7. Known thrombocytopenia < 100.000 platelets/mL 1.8. Prolonged (>20 minutes) or traumatic cardiopulmonar resuscitation (CPR) in the 2 weeks prior to randomization 1.9. History or signs suggesting aortic dissection
2. Cardiogenic shock
3. Estimated door-to-needle time >120 minutes
4. Administration of fibrinolysis in the 14 days prior to randomization
5. Administration of any glycoprotein IIa/IIIb inhibitor in the 24 hours prior to randomization
6. Administration of any Low Molecular Weight Heparin (LMWH) in the 8 hours prior to randomization
7. Actual oral anticoagulant treatment
8. Suspected AMI secondary to occlusion of one lesion treated previously with a percutaneous coronary intervention (within the previous 30 days for angioplasty or conventional stent and within the previous 12 months for coated stents)
9. Dementia or acute confusional state at the time of randomization
10. Subject incapacity or unwillingness to give informed consent -at least, verbally
11. Known renal failure (basal creatinine> 2,5 mg/dl)
12. Reduced life expectancy (<12 months) due to advanced or terminal concomitant condition
13. Subject participation in another clinical trial (assessing a drug or a device) in the 30 days prior to randomization

Diagnostic criteria for the pathologies of the study

Patients with a diagnosis of AMI presenting with:

* Chest pain or any symptom of myocardial ischemia of, at least, 20 minutes of duration, not responding to nitrate therapy and an evolution period of less than 6 hours after symptom onset until randomization process, with, at least, one of the following alterations:
* ST-elevation >=2 mm in 2 or more precordial leads
* ST-elevation >=1 mm in 2 or more anterior leads
* Complete de novo (or probably de novo) left bundle branch block (LBBB)

Estimate of sample size For the following conditions: α = 0.05 (2 tailed), power: 80% (β = 0.20) and assuming a composite event incidence rate (death, reinfarction and disabling CVA) based on previous registries (21.7% in the fibrinolysis group and 12.8% in the PA group), a sample size of 282 patients per group is needed to demonstrate that difference (8.9% in absolute terms and 40% in relative terms). Assuming a loss to follow-up rate of 1%, the total number is 570 patients

Estimated loss of patients prior to randomization During a period of 3 months all patients meeting inclusion criteria who, for any reason, are not enrolled in the study will be included in a registry with an abbreviated CRF recording inclusion/exclusion criteria, the reason for non-enrollment and follow-up at 30 days and 12 months.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Subjects of 75 or more years of age
2. Diagnosis of AMI: chest pain or any symptom of myocardial ischemia of, at least, 20 minutes of duration, not responding to nitrate therapy, an evolution period of less than 6 hours after symptom onset until randomization process, and, at least, one of the following alterations:

   1. ST-elevation >=2 mm in 2 or more precordial leads
   2. ST-elevation >=1 mm in 2 or more anterior leads
   3. Complete de novo (or probably de novo) left bundle branch block (LBBB)
3. Subject should be able to give informed consent prior to randomization process and should agree to fulfill all procedures described in the protocol, including follow-up after hospital discharge. A written consent signed by a close relative with witness is also acceptable.

EXCLUSION CRITERIA:

1. Documented contraindication to the use of fibrinolytics. 1.1. Internal active bleeding or known history of hemorrhagic diathesis 1.2. History of previous CVA of any kind or at any time 1.3. Intracranial tumor, arteriovenous malformation, aneurysm or cerebral aneurysm repair 1.4. Major surgery, parenchymal biopsy, ocular surgery or severe traumatism in the 6 weeks prior to randomization 1.5. Unexplained puncture in a non-compressible vascular location in the last 24 hours prior to randomization 1.6. Confirmed arterial hypertension with a reliable measurement of systolic AP >180 mmHg or diastolic AP >110 mmHg 1.7. Known thrombocytopenia < 100.000 platelets/mL 1.8. Prolonged (>20 minutes) or traumatic cardiopulmonar resuscitation (CPR) in the 2 weeks prior to randomization 1.9. History or signs suggesting aortic dissection
2. Cardiogenic shock
3. Estimated door-to-needle time >120 minutes
4. Administration of fibrinolysis in the 14 days prior to randomization
5. Administration of any glycoprotein IIa/IIIb inhibitor in the 24 hours prior to randomization
6. Administration of any Low Molecular Weight Heparin (LMWH) in the 8 hours prior to randomization
7. Actual oral anticoagulant treatment
8. Suspected AMI secondary to occlusion of one lesion treated previously with a percutaneous coronary intervention (within the previous 30 days for angioplasty or conventional stent and within the previous 12 months for coated stents)
9. Dementia or acute confusional state at the time of randomization
10. Subject incapacity or unwillingness to give informed consent -at least, verbally
11. Known renal failure (basal creatinine> 2,5 mg/dl)
12. Reduced life expectancy (<12 months) due to advanced or terminal concomitant condition
13. Subject participation in another clinical trial (assessing a drug or a device) in the 30 days prior to randomization

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 266 (Actual)
Dates: Start 2005-04; Primary Completion 2008-02 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hector Bueno, MD, PhD, Principal Investigator — Spanish Society of Cardiology (WG on Ischemic Heart Disease and CCUs); Rosa Ana Hernández-Antolín, MD, Principal Investigator — Spanish Society of Cardiology (WG on Interventional Cardiology)
Locations (23):
- Spain (23):
  - Hospital Universitario Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Juan Ramón Jiménez, Huelva, Huelva
  - Complejo Hospitalario Universitario "Juan Canalejo", A Coruña, La Coruña
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Complejo Hospitalario de León, León, León
  - Hospital General Universitario "Gregorio Maranon", Madrid, Madrid
  - Hospital Clínico "San Carlos", Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario "Virgen de la Victoria", Málaga, Málaga
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Complejo Hospitalario de Toledo Hospital Virgen de la Salud, Toledo, Toledo
  - Consorcio Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid
  - Hospital de Cruces, Barakaldo, Vizcaya

REFERENCES:
- [Background] Bardaji A, Bueno H, Fernandez-Ortiz A, Cequier A, Auge JM, Heras M. [Type of treatment and short-term outcome in elderly patients with acute myocardial infarction admitted to hospitals with a primary coronary angioplasty facility. The TRIANA (TRatamiento del Infarto Agudo de miocardio eN Ancianos) Registry]. Rev Esp Cardiol. 2005 Apr;58(4):351-8. Spanish. PMID 15847731
- [Background] Cequier A, Bueno H, Auge JM, Bardaji A, Fernandez-Ortiz A, Heras M. [Characteristics and mortality following primary percutaneous coronary intervention for acute myocardial infarction in Spain. Results from the TRIANA 1 (TRatamiento del Infarto Agudo de miocardio eN Ancianos) Registry]. Rev Esp Cardiol. 2005 Apr;58(4):341-50. Spanish. PMID 15847730
- [Result] Bueno H, Betriu A, Heras M, Alonso JJ, Cequier A, Garcia EJ, Lopez-Sendon JL, Macaya C, Hernandez-Antolin R; TRIANA Investigators. Primary angioplasty vs. fibrinolysis in very old patients with acute myocardial infarction: TRIANA (TRatamiento del Infarto Agudo de miocardio eN Ancianos) randomized trial and pooled analysis with previous studies. Eur Heart J. 2011 Jan;32(1):51-60. doi: 10.1093/eurheartj/ehq375. Epub 2010 Oct 22. PMID 20971744

RESULTS

PARTICIPANT FLOW:
Groups:
- Thrombolysis: Weight adjusted tenecteplase bolus + Unfrationated heparin
  Tenecteplase + UFH (+ clopidogrel, since 01/97)
Period: Overall Study
Arm/Group | Thrombolysis | Primary Angioplasty
Started | 134 | 132
Completed | 132 | 130
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thrombolysis | Primary Angioplasty | Total
Number analyzed (Participants) | 134 | 132 | 266
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 134 | 132 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] — years of age at randomization
  years | 81.0 (4.3) | 81.2 (4.6) | 81.1 (4.5)
Gender [Count of Participants; unit: Participants]
  Female | 76 | 74 | 150
  Male | 58 | 58 | 116
Region of Enrollment [Number; unit: participants]
  Spain | 134 | 132 | 266

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Death or Reinfarction or Disabling Stroke
Description: Incidence of all-cause death or myocardial reinfarction or disabling stroke
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Thrombolysis | Primary Angioplasty
Number analyzed (Participants) | 134 | 132
participants | 34 | 25

2. Primary Outcome: Death/Reinfarction/Disabling Stroke at 30 Days
Description: Incidence of Death or Reinfarction or Disabling Stroke at 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Thrombolysis | Primary Angioplasty
Number analyzed (Participants) | 134 | 132
Participants | 34 | 25
Statistical Analysis 1: Comparison: Thrombolysis vs Primary Angioplasty; Test type: Superiority or Other; p = 0.21, Chi-squared — Unadjusted analysis; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.38 to 1.23]

ADVERSE EVENTS:
Arm/Group | Thrombolysis | Primary Angioplasty
Serious Adverse Events (participants affected / at risk) | 16/134 | 13/132
Other Adverse Events (participants affected / at risk) | 8/134 | 10/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thrombolysis (N=134) | Primary Angioplasty (N=132)
Major bleeding (Blood and lymphatic system disorders) | 5 (5) | 6 (6) — Major haemorrhage
Mechanical complications (Cardiac disorders) | 4 (4) | 4 (4) — Cardiac rupture (free wall rupture, interventiruclar septal rupture, papillary muscle rupture)
Red blood transfusion (Blood and lymphatic system disorders) | 7 (7) | 4 (4)
Major hemorrhage or transfusion (Blood and lymphatic system disorders) | 12 (12) | 9 (9)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thrombolysis (N=134) | Primary Angioplasty (N=132)
Acute renal failure (Renal and urinary disorders) | 8 (8) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No